CLINICAL TRIAL: NCT03970577
Title: Rituximab From the First Episode of Minimal Change Nephrotic Syndrome for Preventing Relapse Risk in Adult Patients: a Multicenter Randomized Controlled Trial
Brief Title: RItuximab From the FIRst Episode of Idiopathic Nephrotic Syndrome
Acronym: RIFIREINS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P170922J; 2018-003437-15 (EudraCT Number)
Record Dates: First submitted 2019-04-15; First posted 2019-05-31 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-04

CONDITIONS: Minimal Change Nephrotic Syndrome (MCNS)
Keywords: Minimal Change Nephrotic syndrome; Rituximab; Relapse rate
MeSH Terms: conditions — Nephrosis, Lipoid | interventions — Rituximab; Prednisone

STUDY DESIGN:
Intervention Model Description: The study will be a single stage phase IIb, randomized, open-label, parallel group, in a 1:1 ratio, active controlled, multicenter trial testing the efficacy and safety of two injections of Rituximab separated by one week (375mg/m2) from initial episode of MCNS in adults.
  The control arm is a standard regimen of oral steroid alone (progressively tapered within 24 weeks).
  At inclusion, all patients will receive oral steroid therapy (Prednisone, 1mg/kg/day, maximum 80 mg/day). For patients without complete remission after 4 weeks of treatment, prednisone will be continued at the same dose until the 8th week. For patients with complete remission after 4 weeks of treatment, doses of prednisone will be progressively reduced between the 4th and the 8th week (0.06 mg/kg by week).
  Patients who reach complete remission by 8 weeks after inclusion will be randomized at this time to receive either Rituximab (experimental group) or the standard steroid regimen (control group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab treatment (Experimental): Two injections of Rituximab (375mg/m2) separated by one week (one at time of randomization and the other one week after) and definitive withdrawal of steroid at the time of second injection of Rituximab (for a total steroids exposure of 9 weeks)
  Interventions: Drug: Rituximab
- Oral steroid treatment (Active Comparator): The patients will continue exclusive oral steroid treatment, that will be progressively tapered, for a total of 24 weeks (by taking into account the initial oral steroid therapy administered during 8 weeks and the oral steroid treatment given after randomization).
  Each patient will be followed up until 18 months after randomization. The patient will have study visits at inclusion, 4 weeks and 8 weeks after inclusion. At the time of randomization, patients who will have reached CR of MCNS will be allocated in test or control group and will be followed up similarly: visits at 1, 4, 16, 24 weeks, 12 and 18 months after randomization.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Rituximab — Two injections of Rituximab (375mg/m2) separated by one week (one at time of randomization and the other one week after) and definitive withdrawal of steroid at the time of second injection of Rituximab (for a total steroids exposure of 9 weeks)
  Other Names: Mabthéra
  Arms: Rituximab treatment
Drug: Prednisone — exclusive oral steroid therapy (progressively tapered with the same procedure for all patients) for a total exposure of 24 weeks (taking into account the initial oral steroid therapy administered during 8 weeks in addition with the oral steroid treatment given after randomization). Each patient will be followed up until 18 months after randomization.
  Other Names: Cortancyl
  Arms: Oral steroid treatment

SUMMARY:
Minimal change nephrotic syndrome (MCNS) is an acquired glomerular disease characterized by massive proteinuria occurring in the absence of glomerular inflammatory lesions or immunoglobulin deposits. MCNS represents a frequent cause of nephrotic syndrome (NS) in adults (10% to 25% of cases). The disease typically takes a chronic course characterized by frequent relapses. Until now, exclusive oral steroid therapy at the dose of 1mg/kg/day (max 80 mg/day) for a minimum of 4 weeks and a maximum of 16 weeks (as tolerated) constitutes the first line treatment of adults with MCNS. Despite of successful remission of initial episode, previous case series showed that 56%-76% of patients experience at least one relapse after steroid-induced remission. The recent MSN trial prospectively showed that 57.9% and 70% of adult patients were in complete remission (CR) after 4 and 8 weeks of oral steroids therapy (1mg/kg/day). Among them, 23.1% of patients displayed at least one relapse episode (after one year-follow-up). Although well tolerated, side effects are common in patients with prolonged and/or repeated courses of steroids and alternative regimens seem highly suitable to reduce the risk of subsequent relapse. Rituximab has recently emerged as a promising therapeutic option in patients with steroids dependent-MCNS. In a multicenter, double-blind, randomized, placebo-controlled trial in children with frequent relapse or with steroid dependent NS, the authors found that the median relapse free period was significantly longer in the Rituximab group than in the placebo group without significant differences concerning serious adverse events. To our knowledge, its use has never been investigated for the initial episode of MCNS with the aim to reduce the subsequent risk of relapse that is a major concern in the management of MCNS patients.

The main objective is to demonstrate, from initial episode of MCNS in adults, once complete remission has occurred, that the use of Rituximab (two injections separated by one week 375mg/m2, with definitive steroids withdrawal after 9 weeks of treatment) may reduce the risk of subsequent MCNS relapse after 12 months of follow-up and may be a safe and an efficient treatment regimen.

The study will be a single stage phase IIb, randomized, open-label, parallel group, in a 1:1 ratio, active controlled, multicenter trial testing the efficacy and safety of two injections of Rituximab separated by one week 375mg/m2 from initial episode of biopsy-proven MCNS in adults. Since Rituximab therapy (when initiated in a context of steroid dependency MCNS) seems to be more effective in patients with complete remission and because of recent data from MSN trial showing that 70% of patients were in complete remission of nephrotic syndrome after 8 weeks of steroids, we decided to maximize the potential benefit, to perform randomization of patients after 8 weeks of steroid treatment. A potential risk factor of relapse is the time of CR occurrence, and because some patients reach CR at 4 weeks and others at 8 weeks, a randomization (1:1) with minimization strategy will be done in order to balance this factor between arms. The primary endpoint will be the incidence of MCNS relapse during the 12 months following randomization defined by the recurrence of nephrotic syndrome (urine protein/creatinine ratio (UPCR) ≥ 300mg/mmol and decreased albumin level (< 30 g/L) in a patient who was in complete remission.

Rituximab is currently considered as an effective therapeutic option to maintain remission in patients with frequently relapsing nephrotic syndrome (FRNS) or steroid-dependent nephrotic syndrome (SDNS). The goal of this prospective study is to determine the potential interest of the use of Rituximab from the initial episode of MCNS to reduce the risk of subsequent relapse, that is a major concern in the management of MCNS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* First episode of Minimal change nephrotic syndrome defined as albumin level < 30 g/L and urine protein/creatinine ratio (UCPR) ≥ 300mg/mmol
* Biopsy-proven MCNS defined on renal biopsy examination by the presence of minimal change glomerular lesions and absence of segmental sclerosis by light microscopy, negative immunofluorescence, or presence of IgM deposits into the mesangium
* Signed informed consent to participate in the study
* Patients who are affiliated with the French health care system

Exclusion Criteria:

Previous administration of Rituximab therapy

* MCNS resulting from a secondary process (lymphoid disorders or malignant disease) or potentially related to treatment known to be associated with MCNS occurrence (Lithium, Interferon, non-steroidal anti-inflammatory drugs)
* Patients with acute infections or chronic active infections
* Positive serological screening test for HIV, B or C hepatitis
* Positive immunological tests for antinuclear and anti-DNA antibodies
* Usual contraindication to steroid or Rituximab
* Immunosuppressed patients, patients with a severe immune deficit
* Patients with hypersensitivity to a monoclonal antibody or biological agents
* Patients with a known allergy to steroid and its excipients or to Rituximab and its excipients or to acetaminophen and its excipients or to cetirizine and its excipients or to protein of murine origin
* Patients with other uncontrolled diseases, including drug or alcohol abuse, severe psychiatric diseases, that could interfere with participation in the trial according to the protocol,
* Patients who have white blood cell count ≤4,000/mm3,
* Patients who have platelet count ≤100,000/mm3,
* Patients who have haemoglobin level <9g/dL,
* Patients who have SGOT or SGPT or bilirubin level greater than 3 times the upper limit of normal
* Patients who have serum creatinine level >150 µmol/l,
* Patients with active cancer or recent cancer (<5 years),
* Females of childbearing potential who don't have an effective method of birth control during the study and during the next 12 months after treatment stop
* Women who are pregnant (positive βHCG at inclusion), or who plan to become pregnant whilst in the trial
* Breastfeeding women
* Severe heart failure (New York Heart Association Class III and IV) or severe, uncontrolled cardiac disease
* Patients who participate simultaneously in another interventional trial
* Patients not willing or able to comply with the protocol requirements
* Patients who are under tutorship or curatorship

Non randomization criteria

* Absence of complete remission after 8 weeks of treatment by steroids (CR is defined as albumin level > 30 g/L and urine protein/creatinine ratio <30mg/mmol ).
* Positive βHCG at randomization (after 8 weeks of treatment by steroids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2023-11-29 (Estimated); Study Completion 2023-11-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of MCNS relapse during the 12 months following randomization | 12 months following randomization
  defined by the recurrence of nephrotic syndrome (urine protein/creatinine ratio (UPCR) ≥ 300mg/mmol and decreased albumin level (< 30 g/L) in a patient who was in complete remission

SECONDARY OUTCOMES:
The relapse rate | 18 months after randomization
  The relapse rate by 18 months of follow-up after randomization
Type of adverse events (AEs) and serious adverse events (SAEs) | 18 months
Frequency of adverse events (AEs) and serious adverse events (SAEs) | 18 months
Severity of adverse events (AEs) and serious adverse events (SAEs) assessed by the CTCAE version 4.0 | 18 months
  The AEs will be recorded by 18 months after randomization and graded according to Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Treatment Burden questionnaire (TBQ) © (Ravaud et al, 2012) | 4 weeks before randomization, 1 week after randomization and 16 weeks after randomization
  The TBQ is a validated questionnaire exploring burden associated with taking medicine, self-monitoring, laboratory exams, medical visits, need for organization, administrative tasks, following advice on diet and physical activity, and social and financial impact of the treatment TBQ is composed of 15 items with rating scale ranging from 0 (best outcome ("not a problem")) to 10 (worst outcome ("large problem")) and an open-ended question. It is unidimensional and a global score (sum of answers to each item) is calculated.
  4 weeks before randomization, 1 week after randomization (i.e. end of treatment for experimental arm) and 16 weeks after randomization (i.e. time of steroids cessation for control arm). The baseline level of treatment burden is assessed at Week -4 (instead of W0 randomization) to avoid a learning bias because the questionnaire would have been administered at time points W0 and W1.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent AUDARD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AUDARD, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION

REFERENCES:
- [Derived] Gauckler P, Matyjek A, Kapsia S, Marinaki S, Quintana LF, Diaz MM, King C, Griffin S, Ramachandran R, Odler B, Eller K, Artan AS, Mirioglu S, Busch M, Schaepe M, Turkmen K, Cheung CK, Pepper RJ, Juarez GF, Pascual J, Aunon P, Garcia-Carro C, Rodriguez A, Alberici F, Luzardo L, Chebotareva N, Schonermarck U, Fernandez L, Radhakrishnan J, Guaman K, Peleg Y, Hoisnard L, Audard V, Papasotiriou M, Krnanska N, Tesar V, Hruskova Z, Bruchfeld A, Stangou M, Lioulios G, Faguer S, Ribes D, Salhi S, Windpessl M, Galesic K, Crnogorac M, Zagorec N, Mayer G, Kronbichler A; RITERM Study Team. Long-Term Outcomes of Rituximab-Treated Adult Patients with Podocytopathies. J Am Soc Nephrol. 2025 Apr 1;36(4):668-678. doi: 10.1681/ASN.0000000520. Epub 2024 Oct 16. PMID 39431468
- [Derived] Christian MT, Maxted AP. Optimizing the corticosteroid dose in steroid-sensitive nephrotic syndrome. Pediatr Nephrol. 2022 Jan;37(1):37-47. doi: 10.1007/s00467-021-04985-1. Epub 2021 Feb 20. PMID 33611671